CLINICAL TRIAL: NCT02073019
Title: A Phase I, Two Part Study Exploring the Safety, Tolerability, Pharmacodynamic and Pharmacokinetic Effect of Ascending Doses of BL-8040 in Healthy Subjects.
Brief Title: A Phase I Study Evaluating Safety, Tolerability, PK and PD of BL-8040 for Stem Cell Mobilization in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BL-8040.02
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Mobilization of Hematopoietic Stem Cells (HSC) to Peripheral Blood (PB)
MeSH Terms: interventions — 4-fluorobenzoyl-TN-14003

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): Each subject will receive a BL-8040 or Placebo on in a randomized double-blind fashion
  Interventions: Drug: BL-8040; Drug: Placebo
- Cohort B (Experimental): Each subject will receive a BL-8040 or Placebo on in a randomized double-blind fashion
  Interventions: Drug: BL-8040; Drug: Placebo
- Cohort C (Experimental): Each subject will receive a BL-8040 or Placebo on in a randomized double-blind fashion
  Interventions: Drug: BL-8040; Drug: Placebo

INTERVENTIONS:
Drug: BL-8040
Drug: Placebo

SUMMARY:
The purpose of this study is to determine whether BL-8040 is safe, tolerable and effective in the mobilization of Hematopoietic Stem Cells (HSC) in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* BMI between 18 and 30 kg/m2 and Weight ≥ 60 Kg
* Subjects must be either surgically sterilized (vasectomy), or if their partner is of childbearing potential, must use two methods of contraception, one of which must be a barrier method, from the first dose until 3 months after the last dose
* Subject is able and willing to comply with the requirements of the protocol

Exclusion Criteria:

* History of clinically significant disease
* Any illness within the 4 weeks prior to the screening examination
* Any history of alcohol and/or drug of abuse addiction and/or active / past (up to 2 years before screening) nicotine consumption
* Clinically relevant deviation from normal in the physical examination and vital signs at screening or baseline
* Clinically relevant laboratory abnormalities identified at screening or baseline
* Positive tests at screening for HIV I & II, hepatitis B and/or hepatitis C in both parts or positive tests for Syphilis, HTLV I & II and Nucleic Acid Test (NAT) for HIV and HBV
* Positive test for urine drugs of abuse or by anamnesis (Barbiturates, Benzodiazepines, Amphetamines, Opiates, Cocaine, Cannabinoids, Methadone, Phencyclidine, and Tricyclic Antidepressants) and/or positive alcohol blood test
* Subjects who have lost or donated in excess of 400 mL of blood within 3 months prior to Day 1 of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | Up to 7 days after treatment comletion

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD, Study Chair — BioLineRx, Ltd.
Locations (1):
- Hadassah Clinical Research Center, Jerusalem, Israel